CLINICAL TRIAL: NCT02966509
Title: Engagement of Patients With Advanced Cancer
Acronym: EPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EPAC1
Record Dates: First submitted 2016-10-10; First posted 2016-11-17 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: End of Life; Advanced Cancer; Lung Neoplasm; Gastric Cancer; Colon Cancer; Glioblastoma Multiforme; Head and Neck Neoplasms; Rectum Cancer; Melanoma; Kidney Cancer; Prostate Cancer; Testicular Neoplasms; Liver Cancer; Cancer of Unknown Origin
MeSH Terms: conditions — Death; Lung Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Glioblastoma; Head and Neck Neoplasms; Rectal Neoplasms; Melanoma; Kidney Neoplasms; Prostatic Neoplasms; Testicular Neoplasms; Liver Neoplasms; Neoplasms, Unknown Primary | interventions — erythromycin propionate-N-acetylcysteinate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Intervention Arm (Experimental): All participants randomized to Arm A will receive the EPAC intervention as well as usual oncologic care.
  Interventions: Behavioral: EPAC
- B: Control Group Arm (No Intervention): All participants randomized to Arm B will receive usual oncologic care.

INTERVENTIONS:
Behavioral: EPAC — Each patient will receive a lay health worker who will engage and educate patients on goals of care documentation and will continue to address goals of care for at least 6 months with patients after enrollment in the study.
  Arms: A: Intervention Arm

SUMMARY:
The Engagement of Patients with Advanced Cancer is an intervention that utilizes well-trained lay health coaches to engage patients and their families in goals of care and shared decision-making after a diagnosis of advanced cancer. Although lay health workers have never been tested in this role, we hypothesize that lay health workers can feasibly improve goals of care documentation and help to reduce unwanted healthcare utilization at the end of life for Veterans diagnosed with new advanced stages of cancer and those diagnosed with recurrent disease.

DETAILED DESCRIPTION:
VAPAHCS proposes to implement and evaluate several critical elements to be in alignment with the VHA's Strategic Goal and priority areas for FY2013. The Engagement of Patients with Advanced Cancer project is an innovative program that will strengthen provider-patient relationship and facilitate whole person care about matters important to Veterans with cancer and important to support network and family. The project is intended to help establish Goals of Care Plan with appropriate documentation, develop, deploy, and evaluate a model of care for persons with cancer that is intended to improve clinical outcomes and experience of care for individuals with advanced cancer who have advanced cancer (stages III, IV or recurrent disease). The intervention provides patients with lay health coaches who assist patients and their families in discussing goals of care and engage in shared-decision making. The goal of the project is to demonstrate that there is improved patient experiences, outcomes, and that the program helps to reduce utilization of health care resources at the end of life.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage III or IV cancer
* Recurrent disease (any stage)
* Ability to consent to study

Exclusion Criteria:

* Patients who are unable to consent to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

REFERENCES:
- [Derived] Patel MI, Agrawal M, Blayney DW, Bundorf MK, Milstein A. Long-Term Engagement of Patients With Advanced Cancer: Results From the EPAC Randomized Clinical Trial. JAMA Oncol. 2024 Jul 1;10(7):905-911. doi: 10.1001/jamaoncol.2024.1221. PMID 38814627
- [Derived] Patel MI, Sundaram V, Desai M, Periyakoil VS, Kahn JS, Bhattacharya J, Asch SM, Milstein A, Bundorf MK. Effect of a Lay Health Worker Intervention on Goals-of-Care Documentation and on Health Care Use, Costs, and Satisfaction Among Patients With Cancer: A Randomized Clinical Trial. JAMA Oncol. 2018 Oct 1;4(10):1359-1366. doi: 10.1001/jamaoncol.2018.2446. PMID 30054634

RESULTS

PARTICIPANT FLOW:
Recruitment Details: August 2013 recruitment for overall study through new patient visit screening, phone calls to patients prior to first oncology appointment, and referral by physicians when diagnosed with recurrent cancers. Recruitment completed in February 2015.
Period: Baseline Satisfaction Survey
Arm/Group | A: Intervention Arm | B: Control Group Arm
Started | 105 | 108
Completed | 101 | 101
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Refused to Answer | 1 | 2
Period: 6 Month Satisfaction Decision Survey
Arm/Group | A: Intervention Arm | B: Control Group Arm
Started | 105 | 108
Completed | 80 | 77
Not Completed | 25 | 31
Not completed — Death | 22 | 25
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Refused to Answer | 0 | 2
Period: 6 Month Satisfaction Survey
Arm/Group | A: Intervention Arm | B: Control Group Arm
Started | 105 | 108
Completed | 58 | 60
Not Completed | 47 | 48
Not completed — Death | 36 | 33
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Refused to Answer | 8 | 11
Period: 6-Month Utilization and Cost
Arm/Group | A: Intervention Arm | B: Control Group Arm
Started | 105 | 108
Completed | 105 | 108
Not Completed | 0 | 0
Period: 15-Month Utilization and Cost
Arm/Group | A: Intervention Arm | B: Control Group Arm
Started | 105 | 108
Completed | 105 | 108
Not Completed | 0 | 0
Period: End of Life Utilization and Cost 6 Month
Arm/Group | A: Intervention Arm | B: Control Group Arm
Started | 105 | 108
Completed | 36 | 33
Not Completed | 69 | 75
Not completed — Patient Still Alive | 69 | 75
Period: End of Life Utilization and Cost 15month
Arm/Group | A: Intervention Arm | B: Control Group Arm
Started | 105 | 108
Completed | 60 | 60
Not Completed | 45 | 48
Not completed — Patient Still Alive | 45 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Intervention Arm | B: Control Group Arm | Total
Number analyzed (Participants) | 105 | 108 | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 36 | 63
  >=65 years | 78 | 72 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (9.20) | 69.4 (9.05) | 69.3 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 103 | 108 | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 99 | 97 | 196
  Unknown or Not Reported | 4 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 4 | 5 | 9
  Black or African American | 5 | 6 | 11
  White | 82 | 83 | 165
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 4 | 9 | 13
Region of Enrollment [Number; unit: participants] — Country
  participants
    United States | 105 | 108 | 213
Cancer Diagnosis [Count of Participants; unit: Participants]
  Thoracic | 41 | 39 | 80
  Gastrointestinal | 26 | 27 | 53
  Genitourinary | 8 | 9 | 17
  Head and Neck | 16 | 15 | 31
  Skin | 7 | 7 | 14
  Other | 7 | 11 | 18
Cancer Stage at Diagnosis [Count of Participants; unit: Participants]
  I | 4 | 3 | 7
  II | 12 | 17 | 29
  III | 30 | 29 | 59
  IV | 59 | 59 | 118
Marital Status [Count of Participants; unit: Participants]
  Married | 35 | 40 | 75
  Unmarried | 70 | 68 | 138
Total Baseline Health Care Costs [Median (Inter-Quartile Range); unit: US Dollars] | 14052 [4613 to 35684] | 11455 [3567 to 29085] | 13090 [4091 to 29729]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Completed Goals of Care Documentation. We Will Evaluate if 75% of Patients in the Intervention Arm Have a Documented Goals of Care Titled Medical Note Within 6 Months of Patient Enrollment in the Study.
Description: Feasibility is defined as at least 75% of patients in the intervention arm with a documented Goals of Care titled medical note within 6 months of patient enrollment in the study.
Time Frame: 6 months after each patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 105 | 108
Participants | 98 | 26

2. Secondary Outcome: Emergency Department Visit (Chart Review)
Description: Emergency Department Use for each patient will be abstracted by electronic medical record chart review for each patient at 6 months after enrollment.
Time Frame: 6 months after patient enrollment
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 105 | 108
visits | 0.74 (1.12) | 0.78 (1.15)

3. Secondary Outcome: Emergency Department Visit (Chart Review)
Description: Emergency Department Use for each patient will be abstracted by electronic medical record chart review for each patient at 15 months after enrollment.
Time Frame: 15 months after patient enrollment
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 105 | 108
Visits | 1.03 (1.40) | 1.20 (1.53)

4. Secondary Outcome: Hospitalization Visits (Chart Review)
Description: Hospitalization use for each patient will be abstracted by electronic medical record chart review for each patient at 6 months after enrollment.
Time Frame: 6 months after patient enrollment
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 105 | 108
Visits | 0.62 (0.80) | 0.56 (0.89)

5. Secondary Outcome: Hospitalization Visits (Chart Review)
Description: Hospitalization use for each patient will be abstracted by electronic medical record chart review for each patient at 15 months after enrollment.
Time Frame: 15 months after patient enrollment
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 105 | 108
Visits | 0.75 (0.94) | 0.88 (1.07)

6. Secondary Outcome: Hospice Referral (Chart Review)
Description: Hospice referral for each patient will be abstracted by electronic medical record chart review for each patient at 6 months after enrollment.
Time Frame: 6 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 105 | 108
Participants | 32 | 16

7. Secondary Outcome: Palliative Care Referral (Chart Review)
Description: Palliative Care Referral for each patient will be abstracted by electronic medical record chart review for each patient at 6 months after enrollment.
Time Frame: 6 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 105 | 108
Participants | 31 | 24

8. Secondary Outcome: Palliative Care Referral (Chart Review)
Description: Palliative Care Referral for each patient will be abstracted by electronic medical record chart review for each patient at 15 months after enrollment.
Time Frame: 15 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 105 | 108
Participants | 31 | 23

9. Secondary Outcome: Change in Patient Satisfaction With Care Using the Consumer Assessment of Health Care Providers and Systems -General Survey
Description: Each patient will receive a satisfaction with care survey (The Consumer Assessment of Health Care Providers and Systems - General (CAHPS)) at baseline and 6 months. We will measure the change in satisfaction from baseline to 6 months. Scores for satisfaction were assessed using the Consumer Assessment of Healthcare Providers and Systems-General survey question #18 which measured rating of health provider, on which scores range from 0 to 10, with higher ratings correspond to higher patient satisfaction. Scores for each group are averaged at baseline and at 6 months.
Time Frame: Change in Patient Satisfaction with Care from baseline to 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 58 | 60
units on a scale | -0.54 (2.40) | -0.99 (2.40)

10. Secondary Outcome: Patient Satisfaction With Decision-Making Using the Satisfaction With Decision Survey
Description: Each patient will receive a validated satisfaction with decision-making survey (The Satisfaction with Decision Survey) at 6 months after study enrollment.Satisfaction with Decision was assessed with the use of the 6-question Satisfaction with Decision Scale, on which scores range from 0 to 5, with higher scores indicating better satisfaction with decision-making. Scores for each group are averaged at 6 months after study enrollment.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A: Intervention Arm | B: Control Group Arm
Number analyzed (Participants) | 80 | 77
units on a scale | 4.73 (0.61) | 4.15 (1.02)

ADVERSE EVENTS:
Time Frame: Time frame for adverse event reporting was at 3, 6, 12, and 15 months
Arm/Group | A: Intervention Arm | B: Control Group Arm
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/108
Other Adverse Events (participants affected / at risk) | 0/105 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No